CLINICAL TRIAL: NCT00656513
Title: A Phase II/III Study Comparing Acupuncture-like Transcutaneous Electrical Nerve Stimulation (ALTENS) Versus Pilocarpine in Treating Early Radiation-Induced Xerostomia
Brief Title: Acupuncture-Like Transcutaneous Electrical Nerve Stimulation (ALTENS) or Pilocarpine in Treating Early Dry Mouth in Patients Undergoing Radiation Therapy for Head and Neck Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RTOG-0537; CDR0000592644
Record Dates: First submitted 2008-04-10; First posted 2008-04-11 (Estimated); Results first posted 2017-08-21 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2017-07

CONDITIONS: Head and Neck Cancer; Xerostomia
Keywords: hypopharyngeal cancer; laryngeal cancer; lip and oral cavity cancer; nasopharyngeal cancer; paranasal sinus and nasal cavity cancer; oropharyngeal cancer; salivary gland cancer; metastatic squamous neck cancer with occult primary; xerostomia; tongue cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Xerostomia; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Nasopharyngeal Neoplasms; Oropharyngeal Neoplasms; Salivary Gland Neoplasms; Tongue Neoplasms | interventions — Pilocarpine

STUDY DESIGN:
Intervention Model Description: One arm Phase II followed by a two-arm Phase III
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pilocarpine: Phase III (Active Comparator)
  Interventions: Drug: Pilocarpine
- ALTENS: Phase III (Experimental)
  Interventions: Procedure: ALTENS
- ALTENS: Phase II (Experimental)
  Interventions: Procedure: ALTENS

INTERVENTIONS:
Drug: Pilocarpine — 5mg by mouth 3 times a day for 12 weeks
  Other Names: pilocarpine hydrochloride
  Arms: Pilocarpine: Phase III
Procedure: ALTENS — Acupuncture-like transcutaneous electrical nerve stimulation (ALTENS) twice weekly for 12 weeks via a Codetron unit
  Other Names: acupuncture-like transcutaneous electrical nerve stimulation
  Arms: ALTENS: Phase II; ALTENS: Phase III

SUMMARY:
RATIONALE: Acupuncture-like transcutaneous electrical nerve stimulation (ALTENS) and pilocarpine may help to relieve chronic xerostomia (dry mouth). It is not yet known which remedy is more effective in treating chronic dry mouth caused by radiation therapy in patients with head and neck cancer.

PURPOSE: This randomized phase II/III trial is studying ALTENS to see how well it works compared with pilocarpine in treating chronic dry mouth caused by radiation therapy in patients with head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility of successfully delivering acupuncture-like transcutaneous electrical nerve stimulation (ALTENS) using the Codetron™ unit in a cooperative group setting in head and neck cancer patients with early radiotherapy-induced xerostomia. (phase II)
* Compare the efficacy of ALTENS treatment vs pilocarpine hydrochloride in these patients in reducing overall xerostomia burden, as measured by the University of Michigan 15-item Xerostomia-Related Quality of Life Scale (XeQOLS) at 9 months after randomization. (phase III)

Secondary

* Evaluate the effect of ALTENS treatment on overall xerostomia burden at 6 months after study entry in these patients. (phase II)
* Compare the efficacy of these treatments in these patients in reducing overall xerostomia burden at 4, 6, and 15 months after randomization. (phase III)
* Compare the efficacy of these treatments in these patients in reducing symptom burden, as measured by the four domains of the XeQOLS (i.e., physical functioning, social functioning, personal/psychological functioning, and pain/discomfort) at 4, 6, 9, and 15 months after randomization. (phase III)
* Compare the efficacy of these treatments in these patients in increasing stimulated (i.e., citric acid primed) whole salivary production (WSP), as measured by sialometry, at 4, 6, 9, and 15 months after randomization. (phase III)
* Compare the efficacy of these treatments in these patients in increasing unstimulated (i.e., basal primed) WSP, as measured by sialometry at 4, 6, 9, and 15 months after randomization. (phase III)
* Compare adverse events associated with these treatments in these patients. (phase III)

OUTLINE: This is a phase II followed by a phase III multicenter study.

* Phase II:Patients undergo placement of surface electrodes at the following acupuncture points: large intestine, spleen, stomach, and conception vessel. Patients then undergo acupuncture-like transcutaneous electrical nerve stimulation (ALTENS) to each of these points using the Codetron™ unit for 20 minutes twice weekly for 12 weeks. No further treatment is given after 12 weeks.
* Phase III:Patients are stratified according to prior use of pilocarpine (no vs yes) and length of time from completion of chemotherapy and/or radiotherapy (3-6 months vs 6-12 months vs > 12 months). Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive oral pilocarpine three times daily for up to 12 weeks in the absence of disease progression or unacceptable toxicity.
  * Arm II: Patients undergo ALTENS treatment using the Codetron™ unit twice weekly for up to 12 weeks in the absence of disease progression or unacceptable toxicity.

Patients undergo quality of life (QOL) assessment at baseline and at 6 months after registration in phase II. In phase III patients complete assessments for basal and stimulated whole salivary production, xerostomia burden, and QOL at baseline and at 4, 6, 9, and 15 months after study entry.

After completion of study therapy, patients are followed at 3 months.

PROJECTED ACCRUAL: A total of 45 patients will be accrued to the phase II portion and 144 patients to the phase III portion of this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of head and neck cancer

  * No clinical evidence of disease recurrence by ear, nose, and throat exam with a nasopharyngeal scope, if indicated, 8 weeks prior to registration
* Completed radiotherapy (i.e., standard or intensity-modulated radiotherapy) with or without chemotherapy ≥ 3 months and up to 2 years prior to study entry

  * Grade 1-2 radiotherapy-induced xerostomia according to the NCI Common Toxicity Criteria for Adverse Effects (CTCAE) v.3.0 and the dry mouth/salivary gland xerostomia scale
  * Must have evidence of residual salivary function with unstimulated (basal) whole salivary production ≥ 0.1 ml/min after having refrained from eating or drinking oral fluid for 2 hours
* No patients with normal saliva production (i.e., no salivary gland changes or no xerostomia)
* No history of serious adverse events after prior treatment with and discontinuation of pilocarpine
* No chronic lymphocytic leukemia

PATIENT CHARACTERISTICS:

* See Disease Characteristics
* Zubrod performance status of 0-2
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other invasive malignancy except non-melanomatous skin cancer or cancer from which the patient has been disease-free for at least 3 years (e.g., carcinoma in situ of the breast, oral cavity, or cervix)
* No concurrent contraindications to pilocarpine (e.g., uncontrolled asthma, miosis, or hypersensitivity)
* No severe, active co-morbidity, including any of the following:

  * Unstable cardiac disease or requirement for a pacemaker in-situ
  * Unstable angina and/or congestive heart failure requiring hospitalization within the past 6 months
  * Transmural myocardial infarction within the past 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days prior to registration
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
* No Sjögren syndrome

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 2 weeks since prior pilocarpine or cevimeline and no concurrent use for ophthalmic or non-ophthalmic indications
* No concurrent regular medications that induce xerostomia (e.g., tricyclic antidepressants, antihistamines with anticholinergic effects, or narcotics)
* No concurrent oral stimulating agents or salivary gland medical stimulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2008-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raimond K. W. Wong, MD, Principal Investigator — Margaret and Charles Juravinski Cancer Centre
Locations (20):
- United States (16):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Hospital of Saint Raphael, New Haven, Connecticut
  - Emory Crawford Long Hospital, Atlanta, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Bloomington Hospital Regional Cancer Institute, Bloomington, Indiana
  - Center for Cancer Care at Goshen General Hospital, Goshen, Indiana
  - Methodist Cancer Center at Methodist Hospital, Indianapolis, Indiana
  - Boston University Cancer Research Center, Boston, Massachusetts
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Schiffler Cancer Center at Wheeling Hospital, Wheeling, West Virginia
- Canada (4):
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
  - McGill Cancer Centre at McGill University, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec

REFERENCES:
- [Result] Wong RK, James JL, Sagar S, Wyatt G, Nguyen-Tan PF, Singh AK, Lukaszczyk B, Cardinale F, Yeh AM, Berk L. Phase 2 results from Radiation Therapy Oncology Group Study 0537: a phase 2/3 study comparing acupuncture-like transcutaneous electrical nerve stimulation versus pilocarpine in treating early radiation-induced xerostomia. Cancer. 2012 Sep 1;118(17):4244-52. doi: 10.1002/cncr.27382. Epub 2012 Jan 17. PMID 22252927
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- ALTENS: Phase II; ALTENS: Phase III: Acupuncture-like transcutaneous electrical nerve stimulation (ALTENS) twice weekly for 12 weeks via a Codetron unit
- Pilocarpine: Phase III: 5mg pilocarpine by mouth 3 times a day for 12 weeks
Period: Overall Study
Arm/Group | ALTENS: Phase II | Pilocarpine: Phase III | ALTENS: Phase III
Started | 48 | 73 | 75
Completed | 44 (Subjects with data available for the primary analysis are considered to have completed the study.) | 43 (Subjects with data available for the primary analysis are considered to have completed the study.) | 53 (Subjects with data available for the primary analysis are considered to have completed the study.)
Not Completed | 4 | 30 | 22
Not completed — Protocol Violation | 1 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 11 | 4
Not completed — Death | 0 | 0 | 1
Not completed — Missing data | 0 | 11 | 9
Not completed — Incomplete treatment | 3 | 0 | 0
Not completed — Treatment completed outside of timeframe | 0 | 3 | 1
Not completed — Missing baseline form | 0 | 5 | 5

BASELINE CHARACTERISTICS:
Population: Eligible patients (i.e. without protocol violation)
Groups:
- Total: Total of all reporting groups
Arm/Group | ALTENS: Phase II | Pilocarpine: Phase III | ALTENS: Phase III | Total
Number analyzed (Participants) | 47 | 73 | 73 | 193
Age, Continuous [Median (Full Range); unit: years] | 60 [24 to 80] | 59 [29 to 78] | 58 [42 to 83] | 58 [24 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 11 | 28
  Male | 40 | 63 | 62 | 165

OUTCOME MEASURES:

1. Primary Outcome: Phase II: Treatment Compliance (Number of Compliant Patients)
Description: Patients completing at least 19 out of 24 ALTENS therapy sessions were categorized as compliant. Fleming's two-stage was used, assuming a successful target compliance rate of 80%, statistical power of 0.87, and a type I error rate of 0.13. If fewer than 9 of the first 13 patients were compliant, then treatment delivery will be deemed not feasible. If there were between 9-12 compliant patients, the second stage analysis would be required to determine feasibility of treatment delivery. If all 13 patients are compliant, treatment delivery will immediately be deemed feasible. The second stage analysis required at least 31 compliant out of 39 overall patients for the treatment delivery to be deemed feasible.
Time Frame: Randomization to 12 weeks
Population: Eligible patients starting protocol treatment
Measure: Count of Participants; unit: Participants
Arm/Group | ALTENS: Phase II
Number analyzed (Participants) | 47
Participants
  First Stage: number analyzed (Participants) | 13
  First Stage | 12
  Second Stage (Overall) | 44

2. Primary Outcome: Phase III: Change From Baseline in Overall Xerostomia Burden at 9 Months
Description: Xerostomia burden is measured by the University of Michigan Xerostomia Related Quality of Life Scale (XeQOLS). The XeQOLS is a validated patient-reported 15-item assessment scale with 4 domains: physical functioning,pain/discomfort, personal/psychologic functioning, and social functioning.The score is the average of all responses of all domains and can range from 0 to 4, with higher scores indicating increased xerostomia burden. Change in xerostomia burden is calculated by subtracting the baseline score from the 9-month score such that a negative change indicates an improvement of the xerostomia burden.
Time Frame: Baseline (randomization) and 9 months
Population: Eligible randomized patients with both baseline and 9 month XeQOLS scores
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Pilocarpine: Phase III | ALTENS: Phase III
Number analyzed (Participants) | 43 | 53
units on a scale | -0.27 [-1.06 to 0] | -0.53 [-0.87 to -0.2]
Statistical Analysis 1: Comparison: Pilocarpine: Phase III vs ALTENS: Phase III; An effect size of 0.50 was chosen for sample size calculation. On the basis of a 2-sided t test with alpha= 0.05 and 1 interim analysis, 130 patients were required for 80% statistical power. Adjustment by 10% for loss to follow-up and retrospective ineligibility of recruited study participants yielded a sample size of 144 patients. Actual power given only 96 patients was 68.6%; Test type: Superiority; p = 0.45, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Phase II: Pecentage of Patients With Beneficial Treatment Response
Description: This secondary objective was to evaluate the effect of ALTENS treatment on overall radiation-induced xerostomia burden by looking at treatment response. Treatment response was determined by a reduction of at least 20% from baseline to 6 months in the University of Michigan Xerostomia Related Quality of Life Scale (XeQOLS). The XeQOLS is a validated patient-reported 15-item assessment scale with 4 domains: physical functioning,pain/discomfort, personal/psychologic functioning, and social functioning.The score is the average of all responses of all domains and can range from 0 to 4. Higher scores indicate increased xerostomia burden. This scale has high reproducibility and sensitivity. For the first and second stage analyses, 4 and 10 patients, respectively, must respond to treatment in order to proceed to the phase III component.
Time Frame: Pre-treatment and 6 months from registration
Population: Eligible patients who started treatment and have both baseline and 6-month XeQOLS scores
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ALTENS: Phase II
Number analyzed (Participants) | 35
percentage of participants | 85.7 [84.9 to 86.5]

4. Secondary Outcome: Change From Baseline in Overall Xerostomia Burden at 4, 6, and 15 Months (Phase III)
Description: as for outcome 2
Time Frame: Baseline, 4, 6, and 15 months from randomization
Population: Eligible patients with both baseline and respective follow-up (4,6,15 months) XeQOLS scores.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Pilocarpine: Phase III | ALTENS: Phase III
Number analyzed (Participants) | 67 | 63
units on a scale
  4 months: number analyzed (Participants) | 67 | 52
  4 months | -0.27 [-0.6 to 0] | -0.47 [-0.8 to -0.13]
  6 months: number analyzed (Participants) | 45 | 47
  6 months | -0.33 [-0.73 to -0.2] | -0.4 [-0.87 to -0.14]
  15 months: number analyzed (Participants) | 67 | 47
  15 months | -0.47 [-0.87 to -0.07] | -0.6 [-1 to -0.2]
Statistical Analysis 1: Comparison: Pilocarpine: Phase III vs ALTENS: Phase III; Test type: Superiority; p = 0.11, Wilcoxon (Mann-Whitney) — Two-sided test of values at 4 months
Statistical Analysis 2: Comparison: Pilocarpine: Phase III vs ALTENS: Phase III; Test type: Superiority; p = 0.31, Wilcoxon (Mann-Whitney) — Two-sided test of values at 6 months
Statistical Analysis 3: Comparison: Pilocarpine: Phase III vs ALTENS: Phase III; Test type: Superiority; p = 0.21, Wilcoxon (Mann-Whitney) — Two-sided test of values at 15 months

5. Secondary Outcome: Change From Baseline in Symptom Burden at 4, 6, 9 and 15 Months (Phase III)
Description: Symptom burden is measured by the University of Michigan Xerostomia Related Quality of Life Scale (XeQOLS). The XeQOLS is a validated patient-reported 15-item assessment scale with 4 domains: physical functioning,pain/discomfort, personal/psychologic functioning, and social functioning. The domain score is the average of all responses on a given domain and can range from 0 to 4, with higher scores indicating increased symptom burden. Change in symptom burden is calculated by subtracting the baseline score from the 9-month score such that a negative change indicates an improvement of the symptom burden.
Time Frame: Baseline, 4, 6, 9 and 15 months from randomization
Population: Eligible patients with both baseline and respective follow-up (4,6, 9,15 months) XeQOLS scores.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Pilocarpine: Phase III | ALTENS: Phase III
Number analyzed (Participants) | 67 | 63
units on a scale
  4-month Physical Functioning: number analyzed (Participants) | 43 | 52
  4-month Physical Functioning | -0.5 [-0.75 to 0] | -0.5 [-0.75 to 0]
  4-month Pain/Discomfort: number analyzed (Participants) | 43 | 52
  4-month Pain/Discomfort | -0.25 [-0.75 to 0] | -0.375 [-1 to 0.125]
  4-month Personal/Psychological Functioning: number analyzed (Participants) | 43 | 52
  4-month Personal/Psychological Functioning | -0.25 [-0.5 to 0.25] | -0.5 [-0.875 to -0.125]
  4-month Social Functioning: number analyzed (Participants) | 43 | 52
  4-month Social Functioning | 0 [-0.67 to 0.33] | -0.33 [-0.835 to 0]
  6-month Physical Functioning: number analyzed (Participants) | 45 | 47
  6-month Physical Functioning | -0.5 [-1 to 0] | -0.5 [-1 to 0]
  6-month Pain/Discomfort: number analyzed (Participants) | 45 | 47
  6-month Pain/Discomfort | -0.25 [-0.5 to 0] | -0.5 [-1 to 0]
  6-month Personal/Psychological Functioning: number analyzed (Participants) | 45 | 47
  6-month Personal/Psychological Functioning | -0.25 [-0.75 to 0] | -0.5 [-1 to -0.25]
  6-month Social Functioning: number analyzed (Participants) | 45 | 47
  6-month Social Functioning | -0.33 [-0.67 to 0.66] | -0.33 [-0.67 to 0]
  9-month Physical Functioning: number analyzed (Participants) | 43 | 53
  9-month Physical Functioning | -0.5 [-1.25 to 0] | -0.5 [-1 to -0.25]
  9-month Pain/Discomfort: number analyzed (Participants) | 43 | 53
  9-month Pain/Discomfort | -0.25 [-0.5 to 0] | -0.5 [-1 to 0]
  9-month Personal/Psychological Functioning: number analyzed (Participants) | 43 | 53
  9-month Personal/Psychological Functioning | -0.5 [-1 to 0.25] | -0.75 [-1 to -0.25]
  9-month Social Functioning: number analyzed (Participants) | 43 | 53
  9-month Social Functioning | -0.66 [-1 to 0.33] | -0.33 [-0.67 to 0]
  15-month Physical Functioning: number analyzed (Participants) | 43 | 47
  15-month Physical Functioning | -0.5 [-1 to 0] | -0.75 [-1.25 to -0.25]
  15-month Pain/Discomfort: number analyzed (Participants) | 43 | 47
  15-month Pain/Discomfort | -0.5 [-1 to 0] | -0.5 [-1 to 0]
  15-month Personal/Psychological Functioning: number analyzed (Participants) | 43 | 47
  15-month Personal/Psychological Functioning | -0.5 [-1 to 0] | -0.75 [-1.25 to -0.25]
  15-month Social Functioning: number analyzed (Participants) | 43 | 47
  15-month Social Functioning | 0 [-1 to 0.33] | -0.33 [-0.67 to 0]
Statistical Analysis 1: Comparison: Pilocarpine: Phase III vs ALTENS: Phase III; Test type: Superiority; p = 0.35, Wilcoxon (Mann-Whitney) — 4-month Physical Functioning score; two-sided test, significance level 0.05
Statistical Analysis 2: Comparison: Pilocarpine: Phase III vs ALTENS: Phase III; Test type: Superiority; p = 0.78, Wilcoxon (Mann-Whitney) — 4 months Pain/Discomfort score; two-sided test, significance level 0.05
Statistical Analysis 3: Comparison: Pilocarpine: Phase III vs ALTENS: Phase III; Test type: Superiority; p = 0.12, Wilcoxon (Mann-Whitney) — 4 months Personal/Psychological Functioning score; two-sided test, significance level 0.05
Statistical Analysis 4: Comparison: Pilocarpine: Phase III vs ALTENS: Phase III; Test type: Superiority; p = 0.28, Wilcoxon (Mann-Whitney) — 4-month Social Functioning score; two-sided test, significance level 0.05
Statistical Analysis 5: Comparison: Pilocarpine: Phase III vs ALTENS: Phase III; Test type: Superiority; p = 0.98, Wilcoxon (Mann-Whitney) — 6-month Physical Functioning score; two-sided test, significance level 0.05
Statistical Analysis 6: Comparison: Pilocarpine: Phase III vs ALTENS: Phase III; Test type: Superiority; p = 0.28, Wilcoxon (Mann-Whitney) — 6-month Pain/Discomfort score; two-sided test, significance level 0.05
Statistical Analysis 7: Comparison: Pilocarpine: Phase III vs ALTENS: Phase III; Test type: Superiority; p = 0.13, Wilcoxon (Mann-Whitney) — 6-month Personal/Psychological Functioning score; two-sided test, significance level 0.05
Statistical Analysis 8: Comparison: Pilocarpine: Phase III vs ALTENS: Phase III; Test type: Superiority; p = 0.58, Wilcoxon (Mann-Whitney) — 6-month Social Functioning score; two-sided test, significance level 0.05
Statistical Analysis 9: Comparison: Pilocarpine: Phase III vs ALTENS: Phase III; Test type: Superiority; p = 0.88, Wilcoxon (Mann-Whitney) — 9-month Physical Functioning score; two-sided test, significance level 0.05
Statistical Analysis 10: Comparison: Pilocarpine: Phase III vs ALTENS: Phase III; Test type: Superiority; p = 0.09, Wilcoxon (Mann-Whitney) — 9-month Pain/Discomfort score; two-sided test, significance level 0.05
Statistical Analysis 11: Comparison: Pilocarpine: Phase III vs ALTENS: Phase III; Test type: Superiority; p = 0.49, Wilcoxon (Mann-Whitney) — 9-month Personal/Psychological Functioning score; two-sided test, significance level 0.05
Statistical Analysis 12: Comparison: Pilocarpine: Phase III vs ALTENS: Phase III; Test type: Superiority; p = 0.45, Wilcoxon (Mann-Whitney) — 9-month Social Functioning score; two-sided test, significance level 0.05
Statistical Analysis 13: Comparison: Pilocarpine: Phase III vs ALTENS: Phase III; Test type: Superiority; p = 0.45, Wilcoxon (Mann-Whitney) — 15-month Physical Functioning; two-sided test, significance level 0.05
Statistical Analysis 14: Comparison: Pilocarpine: Phase III vs ALTENS: Phase III; Test type: Superiority; p = 0.30, Wilcoxon (Mann-Whitney) — 15-month Pain/Discomfort; two-sided test, significance level 0.05
Statistical Analysis 15: Comparison: Pilocarpine: Phase III vs ALTENS: Phase III; Test type: Superiority; p = 0.48, Wilcoxon (Mann-Whitney) — 15-month Personal/Psychological Functioning; two-sided test, significance level 0.05
Statistical Analysis 16: Comparison: Pilocarpine: Phase III vs ALTENS: Phase III; Test type: Superiority; p = 0.68, Wilcoxon (Mann-Whitney) — 15-month Social Functioning; two-sided test, significance level 0.05

6. Secondary Outcome: Change From Baseline in Stimulated Whole Salivary Production (WSP) at 4, 6, 9 and 15 Months (Phase III)
Description: Stimulated (citric acid primed) whole salivary production (WSP) was measured by expectoration weight, with one gram of saliva produced considered as one ml of saliva. WSP is expressed in ml/min calculated by dividing the measured weight or volume of WSP by five. Procedure: Patients refrain from eating, drinking, and smoking at least two hours prior to each measurement. Stimulation is elicited by asking patients to rinse 5 ml of 2% citric acid solution in the mouth for 15 seconds and then completely expectorating the citric acid. For each measurement, patients are asked to expectorate continuously into a pre-weighed dry plastic container over a 5-minute period without swallowing. The collected saliva with the plastic container will be weighed (total weight) immediately after each collection. The total weight minus the weight of the container is the weight or volume of whole saliva collected.
Time Frame: Baseline, 4, 6, 9 and 15 months from randomization
Population: Eligible patients with both baseline and respective follow-up (4,6, 9,15 months) WSP measurements.
Measure: Median (Inter-Quartile Range); unit: ml/min
Arm/Group | Pilocarpine: Phase III | ALTENS: Phase III
Number analyzed (Participants) | 73 | 73
ml/min
  4 months | 0.03 [-0.12 to 1.4] | 0.2 [-0.2 to 0.9]
  6 months | 0.2 [-0.27 to 1.33] | 0.40 [-0.3 to 1.07]
  9 months | 0.99 [0 to 1.9] | 0.60 [-0.17 to 1.44]
  15 months | 0.3 [-0.3 to 1.7] | 0.20 [-0.13 to 2]
Statistical Analysis 1: Comparison: Pilocarpine: Phase III vs ALTENS: Phase III; Test type: Superiority; p = 0.97, Wilcoxon (Mann-Whitney) — 4-month score; two-sided test, significance level 0.05
Statistical Analysis 2: Comparison: Pilocarpine: Phase III vs ALTENS: Phase III; Test type: Superiority; p = 0.83, Wilcoxon (Mann-Whitney) — 6-months; two-sided test, significance level 0.05
Statistical Analysis 3: Comparison: Pilocarpine: Phase III vs ALTENS: Phase III; Test type: Superiority; p = 0.28, Wilcoxon (Mann-Whitney) — 9-months; two-sided test, significance level 0.05
Statistical Analysis 4: Comparison: Pilocarpine: Phase III vs ALTENS: Phase III; Test type: Superiority; p = 0.89, Wilcoxon (Mann-Whitney) — 15-months; two-sided test, significance level 0.05

7. Secondary Outcome: Change From Baseline in Unstimulated Whole Salivary Production (WSP) at 4, 6, 9 and 15 Months (Phase III)
Description: Basal whole salivary production (WSP) was measured by expectoration weight, with one gram of saliva produced considered as one ml of saliva. WSP is expressed in ml/min calculated by dividing the measured weight or volume of WSP by five. Procedure: Patients refrain from eating, drinking, and smoking at least two hours prior to each measurement. For each measurement, patients are asked to expectorate continuously into a pre-weighed dry plastic container over a 5-minute period without swallowing. The collected saliva with the plastic container will be weighed (total weight) immediately after each collection. The total weight minus the weight of the container is the weight or volume of whole saliva collected.
Time Frame: Pre-treatment to 4, 6, 9 and 15 months from randomization
Population: Eligible randomized patients with both baseline and respective follow-up (4,6, 9,15 months) WSP measurements.
Measure: Median (Inter-Quartile Range); unit: ml/min
Arm/Group | Pilocarpine: Phase III | ALTENS: Phase III
Number analyzed (Participants) | 73 | 73
ml/min
  4 months: number analyzed (Participants) | 49 | 63
  4 months | 0 [-0.3 to 0.29] | 0 [-0.28 to 0.38]
  6 months: number analyzed (Participants) | 47 | 58
  6 months | 0 [-0.3 to 0.7] | 0.02 [-0.32 to 0.46]
  9 months: number analyzed (Participants) | 46 | 63
  9 months | 0.056 [-0.1 to 0.9] | 0.04 [-0.2 to 0.587]
  15 months: number analyzed (Participants) | 49 | 57
  15 months | 0.13 [0 to 0.9] | 0.192 [-0.2 to 0.8]
Statistical Analysis 1: Comparison: Pilocarpine: Phase III vs ALTENS: Phase III; Test type: Superiority; p = 0.54, Wilcoxon (Mann-Whitney) — 4-months; two-sided test, significance level 0.05
Statistical Analysis 2: Comparison: Pilocarpine: Phase III vs ALTENS: Phase III; Test type: Superiority; p = 0.99, Wilcoxon (Mann-Whitney) — 6-months; two-sided test, significance level 0.05
Statistical Analysis 3: Comparison: Pilocarpine: Phase III vs ALTENS: Phase III; Test type: Superiority; p = 0.56, Wilcoxon (Mann-Whitney) — 6-months; two-sided test, significance level 0.05
Statistical Analysis 4: Comparison: Pilocarpine: Phase III vs ALTENS: Phase III; Test type: Superiority; p = 0.58, Wilcoxon (Mann-Whitney) — 6-months; two-sided test, significance level 0.05

8. Secondary Outcome: Quality of Life (QOL) as Measured by the University of Washington Head and Neck Questionnaire (UWHNSS) Phase III
Description: The UWHNSS includes ten categories-pain, disfigurement, activity, recreation/entertainment, employment, eating, saliva, taste, speech, mucus/phlegm. Patient scores on the UWHNSS range from 0 to 100 with higher scores indicating declining quality of life. Change in total score was calculated by subtracting baseline from follow-up , thus a positive change score indicates a worsening while a negative change score indicates an improvement.
Time Frame: Baseline and 9 months from randomization.
Population: Eligible randomized patients with both baseline and 9-month UWHNSS total scores.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Pilocarpine: Phase III | ALTENS: Phase III
Number analyzed (Participants) | 43 | 51
units on a scale | -3.64 [-9.09 to 1.82] | -7.27 [-12.73 to -1.81]
Statistical Analysis 1: Comparison: Pilocarpine: Phase III vs ALTENS: Phase III; Test type: Superiority; p = 0.14, t-test, 2 sided — Two-sided test, significance level 0.05

ADVERSE EVENTS:
Description: Adverse events are reported for all eligible patients who started protocol treatment. Subjects experiencing more than one of a given adverse event are counted only once for that adverse event.
Arm/Group | ALTENS: Phase II | Pilocarpine: Phase III | ALTENS: Phase III
Serious Adverse Events (participants affected / at risk) | 1/47 | 0/73 | 1/72
Other Adverse Events (participants affected / at risk) | 7/47 | 51/73 | 27/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ALTENS: Phase II (N=47) | Pilocarpine: Phase III (N=73) | ALTENS: Phase III (N=72)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0
Appendicitis perforated (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ALTENS: Phase II (N=47) | Pilocarpine: Phase III (N=73) | ALTENS: Phase III (N=72)
Tinnitus (Ear and labyrinth disorders) | 0 | 4 | 2
Vision blurred (Eye disorders) | 0 | 5 | 0
Constipation (Gastrointestinal disorders) | 0 | 4 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 5 | 1
Dry mouth (Gastrointestinal disorders) | 5 | 22 | 18
Dysphagia (Gastrointestinal disorders) | 1 | 10 | 9
Chills (General disorders) | 0 | 5 | 0
Fatigue (General disorders) | 1 | 7 | 6
Localized edema [head and neck] (General disorders) | 0 | 1 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 4
Dizziness (Nervous system disorders) | 0 | 5 | 3
Headache (Nervous system disorders) | 0 | 14 | 2
Taste alteration (Nervous system disorders) | 1 | 5 | 4
Insomnia (Psychiatric disorders) | 0 | 4 | 2
Urinary frequency (Renal and urinary disorders) | 0 | 5 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 8 | 2
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 3 | 6
Sweating (Skin and subcutaneous tissue disorders) | 0 | 24 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.